CLINICAL TRIAL: NCT01221246
Title: A Phase 2 Double Blinded, Randomized, Placebo Controlled Dose Escalation Study to Evaluate the Efficacy and the Safety of GM602 in Patients With Acute Middle Cerebral Artery Ischemic Stroke Within an 18-hour Treatment Window
Brief Title: Efficacy and Safety Study of GM602 in Patients With Acute Middle Cerebral Artery Ischemic Stroke Within 18 Hours
Acronym: GMAIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genervon Biopharmaceuticals, LLC (Industry)
Collaborators: University of California, Los Angeles (Other); Huntington Hospital (Other Government); Hoag Memorial Hospital Presbyterian (Other); Columbia University (Other); California Pacific Medical Center Research Institute (Other); University Hospital Erlangen (Other); Sarasota Memorial Hospital (Other); University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEN-002
Record Dates: First submitted 2010-10-11; First posted 2010-10-14 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Stroke
Keywords: Acute Middle Cerebral Artery Ischemic Stroke within 18 hours
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GM602 (Experimental): First 9 moderate patients (either co-treated or not co-treated) will be randomized to receive 320 mg/dose of GM602 or placebo in a 2:1 ratio, then the next 9 moderate patients (either co-treated or not co-treated) will be randomized to receive 480 mg/dose of GM602 or placebo in a 2:1 ratio. Concurrently, 18 severe patients will be randomized in the same manner. Total 12 moderate and 12 severe patients will receive GM602.
  Interventions: Drug: GM602
- Placebo Comparator (Placebo Comparator): First 9 moderate patients (either co-treated or not co-treated) will be randomized to receive 320 mg/dose of GM602 or placebo in a 2:1 ratio; then the next 9 moderate patients (either co-treated or not co-treated) will be randomized to receive 480 mg/dose of GM602 or placebo in a 2:1 ratio. Concurrently, 18 severe patients will be randomized in the same manner. Total 6 moderate and 6 severe patients receive Placebo.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: GM602 — First 9 moderate patients (either co-treated or not co-treated) will be randomized to receive 320 mg/dose of GM602 or placebo in a 2:1 ratio, then the next 9 moderate patients (either co-treated or not co-treated) will be randomized to receive 480 mg/dose of GM602 or placebo in a 2:1 ratio. Concurrently, 18 severe patients will be randomized in the same manner. Total 12 moderate and 12 severe patients will receive GM602.
  Other Names: GM6; GM604; GM608; MNTF
  Arms: GM602
Drug: Placebo Comparator — First 9 moderate patients (either co-treated or not co-treated) will be randomized to receive 320 mg/dose of GM602 or Matching Placebo (Bacteriostatic Saline) for GM602 in a 2:1 ratio, then the next 9 moderate patients (either co-treated or not co-treated) will be randomized to receive 480 mg/dose of GM602 or placebo in a 2:1 ratio. Concurrently, 18 severe patients will be randomized in the same manner. Total 6 moderate and 6 severe patients will receive placebo.
  Other Names: Bacteriostatic saline
  Arms: Placebo Comparator

SUMMARY:
The purpose of this research study is to determine whether the investigational drug GM602, is effective and safe in the treatment of ischemic stroke (strokes caused by a blood clot blocking the flow of blood through one, or more of the blood vessels supplying the brain) when administered up to 18 hours after symptoms begin.

DETAILED DESCRIPTION:
Stroke is a serious and life threatening disease. About 85% of all strokes are ischemic, caused by a blood clot or plaque that blocks a blood vessel in the brain. The thrombolytic drug tissue plasminogen activator (tPA) is the only early treatment for acute ischemic stroke approved by the FDA. Treatment with tPA must be administered within three hours of the stroke onset. Furthermore, tPA treatment carries a recognized risk of bleeding in the brain. GM602 is an investigational drug that may act as a neuroprotectant in patients who have had a stroke. It is thought to stop cell death and reduce inflammation in the injured area of the brain. This study is designed to evaluate the safety and efficacy of GM602 administered intravenously to patients in three consecutive daily doses of 320 mg/dose or 480 mg/dose, the initial dose administered within 18 hours after onset of acute ischemic stroke in the Middle Cerebral artery region.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Be eligible for MRI or CT scan
* Have suffered acute ischemic stroke in the middle cerebral artery (MCA) distribution, as verified by the Screening diffusion-weighted imaging (DWI) abnormality and Screening perfusion-weighted imaging pressure-work index (PWI ) abnormality
* Have NIH Stroke Scale (NIHSS) score total score of 9-20 inclusive at screening
* Have suffered acute ischemic stroke within 18 hours
* Have been functionally independent with a Modified Rankin Score (mRS) of 0 or 1 prior to suffering stroke
* Patients who received tPA or FDA approved mechanical device can also enroll
* completed informed consent form

Exclusion Criteria:

* Have history of stroke in the past 3 months
* Cannot be evaluated using MRI/CT
* Have stroke of the brainstem or cerebellum
* Have clinical presentation consistent with acute MI by EKG criteria (STEMI) at screening
* Have hemorrhage revealed by CT or MRI scan
* Have > 1/3 MCA territory HYPER intensity as seen on MRI OR >1/3 MCA territory HYPO intensity as seen on CT
* Have blood sugar level >400 mg/DL or<50 mg/dL
* Have kidney disease, creatinine > 2.0
* Have had recent (within 90 days) serious head trauma or head trauma with loss of consciousness
* Have any prior history of seizure
* Have clinically relevant pre-existing neurological deficit (Historical Rankin score ≥ 2)
* Have any other known clinically significant medical disorder (cardiovascular, hepatic, renal, endocrine, respiratory, immunological, cancer, AIDS)
* Life expectancy of less than 6 months due to comorbid conditions
* Women of child bearing potential who are pregnant or breast-feeding or unable to practice birth control during the study period
* Have participated in any other trial of an investigational agent within 90 days prior to screening
* Informed consent cannot be obtained
* Unable to participate in study visits

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-03-08 (Actual); Primary Completion 2016-07-07 (Actual); Study Completion 2016-07-07 (Actual)

PRIMARY OUTCOMES:
Functional Outcome as measured by the difference in percent change in NIHSS from baseline to 90 days in patients treated with GM602 within 18 hours compared to treated with placebo as primary efficacy endpoint | Day 90
  NIH Stroke Scale is a standardized neurological examination intended to describe the neurological deficits found in large groups of stroke patients participating in treatment trials. Percent change from baseline in NIHSS is calculated and compared.

SECONDARY OUTCOMES:
Functional Outcome as measured by the difference in percent change in NIHSS from baseline to 30 days in patients treated with GM602 compared to treated with placebo | Day 30
  Percent change in NIHSS from baseline to 30 days in patients treated with any active dose of GM602 compared with placebo
Percent change in Barthel Index (BI) from baseline to 90 days in patients treated with GM602 compared to treated with placebo | Day 90
  The Barthel Index is measured using both historical and direct observational information. It measures self-care and mobility and will help define the degree of residual disability. Percent change from baseline in BI is calculated.
Percent change in Barthel Index (BI) from baseline to 30 days in patients treated with GM602 compared to treated with placebo | Day 30
  Percent change in BI from baseline to 30 days in patients treated with any active dose of GM602 compared with placebo
Proportion of patients treated with any active dose of GM602 compared with placebo at each mRS level at 90 days | Day 90
  compared with placebo at each modified Rankin Scale (mRS) level at 90 days.
Proportion of patients treated with any active dose of GM602 compared with placebo at each mRS level at 30 days | Day 30
  compared with placebo at each modified Rankin Scale (mRS) level at 30 days.
Secondary safety endpoint as measured by all cause mortality data through 3 months for patients treated with GM602 compared with placebo | Day 90
  all cause mortality data through 3 months

OTHER OUTCOMES:
Primary Safety Endpoints | througyh 3 months
  Adverse events, Fatal intracranial hemorrhage (ICH). nonfatal symptomatic parenchymal hemorrhage, or other symptomatic ICH, Neurological deterioration during hospitalization, Number of seizures after stroke, Respiratory compromise as observed by respiratory rate

CONTACTS AND LOCATIONS:
Overall Officials: Arbi G Ohanian, MD, Principal Investigator — Huntington Memorial Hospital; Sidney Starkman, MD, Principal Investigator — UCLA Stroke Center; Jeff Saver, MD, Principal Investigator — UCLA Stroke Center; David Brown, MD, Principal Investigator — Hoag Memorial Hospital Presbyterian; Stephan A Mayer, M.D., Principal Investigator — Columbia University; Nobl Barazangi, M.D., Principal Investigator — California Pacific Medical Center Research Institute; Thomas G Devlin, M.D., Principal Investigator — University Erlanger Hospital; Mauricio Concha, M.D., Principal Investigator — Sarasota Memorial Hospital; Anand Vaishnav, M.D., Principal Investigator — University of Louisville
Locations (8):
- United States (8):
  - UCLA Stroke Center (Departments of Emergency Medicine and Neurology at the University of California, Los Angeles Medical Center), Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Huntington Memorial Hospital Stroke Center, Pasadena, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of Louisville, Louisville, Kentucky
  - Columbia University Medical Center, New York, New York
  - University Erlanger Hospital, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No